CLINICAL TRIAL: NCT04937244
Title: Pilot Study Evaluating the Optimization of the ORBEYE Blue Light Filter During Fluorescence-Guided Resection of Gliomas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Collaborators: Olympus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2021-SE-01
Record Dates: First submitted 2021-06-08; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Malignant Glioma of Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with new or recurrent malignant gliomas (Experimental)
  Interventions: Diagnostic Test: 5ALA exoscopic fluorescence filter

INTERVENTIONS:
Diagnostic Test: 5ALA exoscopic fluorescence filter — Visualization of tumor tissue with 5ALA will be done in the operating room to localize neoplastic tissue. The operation will be conducted in a standard fashion uninfluenced by the imaging on the ORBEYE exoscope. The ORBEYE exoscope will be used with the blue light filter after tacking up dura upon first visualization of tumor tissue prior to direct resection. Images will be taken prior to, during and at the end of the planned resection. The ORBEYE exoscope will be set up at constant distances from the target and incident light intensities. The focal distance and light intensity settings will be recorded from the data displayed on the microscope. The ORBEYE exoscope or standard operating microscope (depending on surgeon preference) will then be used in the standard fashion of an operative microscope with a fluorescent filter, to assist with surgical resection as per the surgeon's preference. Resection will proceed according to current standard of care.

SUMMARY:
Fluorescence-guided resection using 5-ALA induced tumor fluorescence of malignant gliomas allows for better identification of tumor tissue and more radical resection in select patients and improvements in progression-free and overall survival. With new developments in surgical microscopy, the development of digital exoscopes have provided advanced visualization as well as improvements in ergonomics and accessibility of the surgical field. The use of the exoscope in 5-ALA fluorescence-guided tumor surgery has the potential to enhance the ability of the surgeon to remove brain tumors with high efficacy. While algorithms for use of 5-ALA fluorescence have been optimized for use with traditional microscopes, the use of fluorescence techniques in newer digital exoscopes have not been developed. The primary outcome of the study is to obtain parameters to optimize visualization of fluorescence intensity and perform optimization based on the intensities achieved. The operating ORBEYE exoscope will be fitted with a blue light filter. All experiments will be performed in darkened operating rooms. The ORBEYE exoscope will be set up at constant distances from the target and incident light intensities. The focal distance and light intensity settings will be recorded from the data displayed on the microscope. Patients (experimental group) will receive 5ALA treatment before operation, blue light filter imagining will take place after tacking up dura and prior to direct resection. The expected outcomes of image analysis will be to have a set of exoscope parameters optimized for visualization of 5ALA tissue in different tumor types. This 5ALA characterization of visualization parameters has never been completed on an exoscope. Optimizing ORBEYE exoscope parameters will define a standard in glioma resection using 5ALA under a novel exoscopic filter as well as contribute insight into the use of the fluorescent filter for additional tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥ 18 years of age
* Must have a suspected or biopsy-proven glioma (World Health Organization grade II or IV), new or recurrent
* Indication for craniotomy for removal of a suspected or recurrent brain tumor
* Karnofsky Performance Scale ≥ 60%
* Willing and able to provide informed consent or have surrogate consent by legally authorized representative

Exclusion Criteria:

* Male and female < 18 years of age
* Porphyria, hypersensitivity to porphyrins
* Renal insufficiency as defined by a creatinine > 2.0 mg/dL
* Hepatic insufficiency as diagnosed in preoperative medical clearance evaluation
* Females of childbearing potential with a positive pregnancy test
* Nursing women
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-05-11 (Estimated); Study Completion 2022-05-11 (Estimated)

PRIMARY OUTCOMES:
Focal Distance | 6 weeks
  To characterize optimal focal distance on the 5ALA fluorescence ORBEYE exoscope microscope during glioma removal
Light Intensity | 6 weeks
  To characterize optimal light intensity settings on the 5ALA fluorescence ORBEYE exoscope microscope during glioma removal
Working Angle | 6 weeks
  To characterize optimal working angle position on the 5ALA fluorescence ORBEYE exoscope microscope during glioma removal

SECONDARY OUTCOMES:
Usability of 5ALA exoscope filter as assessed by overall surgery length | 6 weeks
  To determine functionality and performance reliability of the blue light excitation filter on the ORBEYE exoscope platform with overall surgery length
Usability of 5ALA exoscope filter as assessed by surgeon qualitative assessment | 6 weeks
  To determine functionality and performance reliability of the blue light excitation filter on the ORBEYE exoscope platform with surgeon qualitative assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belykh E, Miller EJ, Patel AA, Bozkurt B, Yagmurlu K, Robinson TR, Nakaji P, Spetzler RF, Lawton MT, Nelson LY, Seibel EJ, Preul MC. Optical Characterization of Neurosurgical Operating Microscopes: Quantitative Fluorescence and Assessment of PpIX Photobleaching. Sci Rep. 2018 Aug 22;8(1):12543. doi: 10.1038/s41598-018-30247-6. PMID 30135440
- [Background] Langer DJ, White TG, Schulder M, Boockvar JA, Labib M, Lawton MT. Advances in Intraoperative Optics: A Brief Review of Current Exoscope Platforms. Oper Neurosurg. 2020 Jul 1;19(1):84-93. doi: 10.1093/ons/opz276. PMID 31529083
- [Background] Hadjipanayis CG, Widhalm G, Stummer W. What is the Surgical Benefit of Utilizing 5-Aminolevulinic Acid for Fluorescence-Guided Surgery of Malignant Gliomas? Neurosurgery. 2015 Nov;77(5):663-73. doi: 10.1227/NEU.0000000000000929. PMID 26308630